CLINICAL TRIAL: NCT01089725
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE.
Brief Title: Efficacy And Safety Study Of Tanezumab Subcutaneous Administration In Osteoarthritis - A Subcutaneous/Intravenous Bridging Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091027; SC/IV OA STUDY (Other: Alias Study Number)
Record Dates: First submitted 2010-03-11; First posted 2010-03-18 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis; Arthritis; Pain
Keywords: safety; efficacy; parallel group; double-blind; multicenter; injection; infusion; osteoarthritis; bridging; subcutaneous; intravenous; tanezumab
MeSH Terms: conditions — Osteoarthritis; Arthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo IV; Biological: Placebo SC
- 2.5 mg tanezumab SC and placebo IV (Experimental)
  Interventions: Biological: Tanezumab SC; Biological: Placebo IV
- 5 mg tanezumab SC and placebo IV (Experimental)
  Interventions: Biological: Tanezumab SC; Biological: Placebo IV
- 10 mg tanezumab SC and placebo IV (Experimental)
  Interventions: Biological: Tanezumab SC; Biological: Placebo IV
- 10 mg tanezumab IV (Experimental)
  Interventions: Biological: Tanezumab IV; Biological: Placebo SC

INTERVENTIONS:
Biological: Placebo IV — 1 ml of placebo administered SC and IV once every 8 weeks.
  Arms: Placebo
Biological: Placebo SC — 1 ml of placebo administered SC and IV once every 8 weeks.
  Arms: Placebo
Biological: Tanezumab SC — 1 ml tanezumab injection SC administered every 8 weeks
  Arms: 2.5 mg tanezumab SC and placebo IV
Biological: Placebo IV — 1 ml placebo administered IV every 8 weeks
  Arms: 2.5 mg tanezumab SC and placebo IV
Biological: Tanezumab SC — 1 ml tanezumab injection SC administered every 8 weeks
  Arms: 5 mg tanezumab SC and placebo IV
Biological: Placebo IV — 1ml placebo administered IV every 8 weeks
  Arms: 5 mg tanezumab SC and placebo IV
Biological: Tanezumab SC — 1 ml tanezumab injection SC administered every 8 weeks
  Arms: 10 mg tanezumab SC and placebo IV
Biological: Placebo IV — 1ml placebo administered IV every 8 weeks
  Arms: 10 mg tanezumab SC and placebo IV
Biological: Tanezumab IV — 1 ml tanezumab injection IV administered every 8 weeks
  Arms: 10 mg tanezumab IV
Biological: Placebo SC — 1ml placebo administered SC every 8 weeks
  Arms: 10 mg tanezumab IV

SUMMARY:
This is an efficacy and safety study of 3 doses (2.5 mg, 5 mg and 10mg) of tanezumab administered subcutaneously versus placebo. This study will also compare a subcutaneous (SC) administration of 10 mg of tanezumab) with an intravenous (IV) administration of 10 mg of tanezumab. Each person will receive an IV infusion and a SC infusion. The study will last 16 weeks for those who wish to enter a 64-week extension study or 24 weeks for those who do not.

DETAILED DESCRIPTION:
This study was terminated on 08 Nov 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis (OA) of the knee according to American College of Rheumatology (ACR) criteria with a Kellgren- Lawrence score of greater than or equal to 2
* 18 years of age or greater
* Two methods of birth control one of which must be barrier if of childbearing potential
* Willing to discontinue pain medication except as permitted per protocol

Exclusion Criteria:

* Pregnancy or wishing to be pregnant during the course of the study, lactating women
* Body Mass Index (BMI) greater than 39
* Clinically significant cardiac, neurological, psychiatric conditions and other conditions that are excluded by the protocol.
* Previous exposure to a Nerve Growth Factor (NGF) antibody

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2010-03-30 (Actual); Primary Completion 2010-11-08 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (89):
- United States (89):
  - Vaughn H. Mancha, Jr., MD, PC, Montgomery, Alabama
  - Novara Clinical Research, Mesa, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - West Coast Radiology Center, Anaheim, California
  - Providence Clinical Research, Burbank, California
  - Valley Research, Fresno, California
  - Allergy and Rheumatology Medical Clinic, Inc., La Jolla, California
  - Triwest Research Associates, La Mesa, California
  - Synergy Clinical Research Center, National City, California
  - Benchmark Research, Sacramento, California
  - Probe Clinical Research Corp., Santa Ana, California
  - Trinity Clinical Trials, Santa Ana, California
  - FMC Clinical Trials, Upland, California
  - Colorado Hematology, Englewood, Colorado
  - Colorado Orthopedic Consultants, P.C., Englewood, Colorado
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Office of Cynthia Morgan, MD, Washington D.C., District of Columbia
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - BayCare Outpatient Imaging at Bardmoor, Largo, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - St. Petersburg Arthritis Center, St. Petersburg, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Sonoma Clinical Research, LLC., Boise, Idaho
  - Sonora Clinical Research, Boise, Idaho
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Wichita Clinic PA, Wichita, Kansas
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - BenchMark Research, Metairie, Louisiana
  - Arthritis Treatment Center, Frederick, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Ann Arbor Clinical Reserch, Ann Arbor, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - Arthritis Associates, PLLC, Hattiesburg, Mississippi
  - Billings Clinic Infusion Center, Billings, Montana
  - Billings Clinic Research Center, Billings, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Midwest Minor Medical, Omaha, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - Andrew Porges, MD, PC, Roslyn, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Greensboro Imaging, Greensboro, North Carolina
  - Pharmquest, Greensboro, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - LION Research, Norman, Oklahoma
  - McBride Clinic, Norman, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Lebanon Internal Medicine Associates, Lebanon, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, LLP, Wyomissing, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - SoFHA Clinical Research, Johnson City, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - Westbury Medical Clinic, Houston, Texas
  - Asif Cochinwala, MD, P.A., Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Little York Medical Center, Houston, Texas
  - Internist Associates of Texas, Kingwood, Texas
  - Accurate Clinical Research Inc, Nassau Bay, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Benchmark Research, San Angelo, Texas
  - Pioneer Research Solutions, Inc, Sugar Land, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Hypothe Test, LLC, Roanoke, Virginia
  - Mountain State Clinical Research, Clarksburg, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Brown MT, Cornblath DR, Koltzenburg M, Gorson KC, Hickman A, Pixton GC, Gaitonde P, Viktrup L, West CR. Peripheral Nerve Safety of Nerve Growth Factor Inhibition by Tanezumab: Pooled Analyses of Phase III Clinical Studies in Over 5000 Patients with Osteoarthritis. Clin Drug Investig. 2023 Jul;43(7):551-563. doi: 10.1007/s40261-023-01286-3. Epub 2023 Jul 18. PMID 37460782
- [Derived] Berenbaum F, Schnitzer T, Kivitz A, Viktrup L, Johnston E, Yang R, Whalen E, Tive L, Semel D. Gender, age, disease severity, body mass index and diabetes may not affect response to subcutaneous tanezumab in patients with osteoarthritis after 16 weeks of treatment. A subgroup analysis of placebo-controlled trials. Int J Clin Pract. 2021 Dec;75(12):e14975. doi: 10.1111/ijcp.14975. Epub 2021 Oct 21. PMID 34626502
- [Derived] Berenbaum F, Schnitzer TJ, Kivitz AJ, Viktrup L, Hickman A, Pixton G, Brown MT, Davignon I, West CR. General Safety and Tolerability of Subcutaneous Tanezumab for Osteoarthritis: A Pooled Analysis of Three Randomized, Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2022 Jun;74(6):918-928. doi: 10.1002/acr.24637. Epub 2022 Mar 25. PMID 33973384
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091027&StudyName=Efficacy%20And%20Safety%20Study%20Of%20Tanezumab%20Subcutaneous%20Administration%20In%20Osteoarthritis%20-%20A%20Subcutaneous/Intravenous%20Bridging%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) subcutaneous injection along with placebo matched to tanezumab intravenous infusion at Baseline and Week 8.
- Tanezumab 2.5 mg Subcutaneous Injection: Tanezumab (RN624 or PF-04383119) 2.5 milligram (mg) subcutaneous injection along with placebo matched to tanezumab intravenous infusion at Baseline and Week 8.
- Tanezumab 5 mg Subcutaneous Injection: Tanezumab (RN624 or PF-04383119) 5 mg subcutaneous injection along with placebo matched to tanezumab intravenous infusion at Baseline and Week 8.
- Tanezumab 10 mg Subcutaneous Injection: Tanezumab (RN624 or PF-04383119) 10 mg subcutaneous injection along with placebo matched to tanezumab intravenous infusion at Baseline and Week 8.
- Tanezumab 10 mg Intravenous Infusion: Tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion along with placebo matched to tanezumab subcutaneous injection at Baseline and Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Started | 72 | 75 | 65 | 87 | 86
Treated | 72 | 74 | 63 | 86 | 84
Completed | 6 | 7 | 4 | 8 | 6
Not Completed | 66 | 68 | 61 | 79 | 80
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 4 | 3 | 1 | 0 | 4
Not completed — Lost to Follow-up | 2 | 2 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 4 | 5 | 4
Not completed — Study Terminated by Sponsor | 51 | 56 | 53 | 68 | 68
Not completed — Randomized, but not treated | 0 | 1 | 2 | 1 | 2
Not completed — Other | 3 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion | Total
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84 | 379
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 8 | 3 | 7 | 4 | 3 | 25
  45 to 64 years | 38 | 48 | 32 | 62 | 56 | 236
  Greater than or equal to (>=) 65 years | 26 | 23 | 24 | 20 | 25 | 118
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 36 | 54 | 48 | 233
  Male | 25 | 26 | 27 | 32 | 36 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Baseline, Week 16
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Baseline | 7.31 (1.41) | 7.70 (1.46) | 7.48 (1.43) | 7.51 (1.29) | 7.24 (1.37)
  Change at Week 16 | -2.79 (2.14) | -3.84 (2.79) | -3.77 (2.62) | -3.88 (2.72) | -3.63 (2.41)

2. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 16
Description: The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in the index joint in the past 48 hours. It is calculated as the mean of the scores from the 17 individual questions scored on a NRS of 0 to 10, where higher scores indicate worse function. Total score range for WOMAC physical function subscale score is 0 to 10, where higher scores indicate worse function.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). LOCF method was used to impute missing values.. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 83
units on a scale
  Baseline | 6.99 (1.67) | 7.25 (1.60) | 7.03 (1.64) | 7.12 (1.42) | 6.75 (1.42)
  Change at Week 16 | -2.29 (2.02) | -3.28 (2.89) | -3.22 (2.49) | -3.51 (2.57) | -3.18 (2.28)

3. Primary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Osteoarthritis Score at Week 16
Description: Participants answered the question: "Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (severe symptoms and inability to carry out most normal activities) and 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated severe condition.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). LOCF method was used to impute missing values. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 83
units on a scale
  Baseline | 3.47 (0.63) | 3.43 (0.64) | 3.43 (0.61) | 3.49 (0.65) | 3.30 (0.51)
  Change at Week 16 | -0.81 (0.87) | -1.03 (1.02) | -0.92 (0.92) | -1.08 (1.10) | -0.92 (0.97)

4. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale at Weeks 1, 2, 4, 8, and 12
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Change at Week 1 | -2.15 (2.25) | -3.06 (2.47) | -2.67 (2.56) | -3.27 (2.49) | -3.41 (2.76)
  Change at Week 2 | -2.46 (2.28) | -3.76 (2.69) | -3.23 (2.70) | -3.19 (2.67) | -2.59 (2.64)
  Change at Week 4 | -2.74 (2.20) | -4.15 (2.72) | -3.63 (2.59) | -3.89 (2.83) | -3.58 (2.47)
  Change at Week 8 | -2.74 (2.09) | -3.89 (2.76) | -3.80 (2.64) | -3.89 (2.73) | -3.59 (2.38)
  Change at Week 12 | -2.81 (2.13) | -3.87 (2.76) | -3.81 (2.67) | -3.88 (2.72) | -3.62 (2.42)

5. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale at Weeks 1, 2, 4, 8, and 12
Description: as for outcome 2
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). LOCF method was used to impute missing values. Here 'overall number of participants analyzed' signifies those who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 83
units on a scale
  Change at Week 1 | -1.75 (2.24) | -2.78 (2.49) | -2.22 (2.26) | -2.99 (2.30) | -2.99 (2.46)
  Change at Week 2 | -1.97 (2.08) | -3.27 (2.73) | -2.89 (2.57) | -3.01 (2.46) | -2.45 (2.36)
  Change at Week 4 | -2.21 (2.07) | -3.55 (2.81) | -3.20 (2.52) | -3.57 (2.53) | -3.17 (2.31)
  Change at Week 8 | -2.26 (2.01) | -3.31 (2.86) | -3.28 (2.53) | -3.51 (2.58) | -3.13 (2.25)
  Change at Week 12 | -2.31 (2.02) | -3.29 (2.87) | -3.27 (2.55) | -3.50 (2.58) | -3.16 (2.29)

6. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Weeks 1, 2, 4, 8, and 12
Description: as for outcome 3
Time Frame: Baseline, Weeks 1, 2, 4, 8, and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 83
units on a scale
  Change at Week 1 | -0.57 (0.82) | -0.82 (0.94) | -0.75 (0.86) | -0.87 (0.85) | -0.88 (1.04)
  Change at Week 2 | -0.67 (0.86) | -0.93 (1.05) | -0.83 (0.89) | -0.94 (1.01) | -0.58 (0.93)
  Change at Week 4 | -0.76 (0.76) | -1.12 (1.03) | -1.02 (0.92) | -1.03 (1.10) | -0.88 (0.90)
  Change at Week 8 | -0.78 (0.83) | -1.07 (1.00) | 0.95 (0.92) | -1.08 (1.10) | -0.90 (0.96)
  Change at Week 12 | -0.81 (0.87) | -1.05 (0.99) | -0.94 (0.93) | -1.08 (1.10) | -0.92 (0.97)

7. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: The OMERACT-OARSI responder index is based on 3 parameters. OMERACT-OARSI response: greater than or equal to (>=) 50 percent (%) improvement from baseline and absolute change from baseline of >=2 units at week of interest in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score range: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score range: 0-10, higher score=higher pain/difficulty).
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
percentage of participants
  Week 1 | 41.7 | 68.9 | 58.7 | 68.6 | 64.3
  Week 2 | 54.2 | 68.9 | 68.3 | 64.0 | 59.5
  Week 4 | 63.9 | 78.4 | 74.6 | 72.1 | 73.8
  Week 8 | 59.7 | 74.3 | 74.6 | 79.1 | 76.2
  Week 12 | 61.1 | 74.3 | 74.6 | 79.1 | 76.2
  Week 16 | 61.1 | 74.3 | 74.6 | 79.1 | 76.2

8. Secondary Outcome: Percentage of Participants With at Least 30%, 50%, 70% and 90% Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: as for outcome 1
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
percentage of participants
  Week 1: >=30% reduction | 36.1 | 54.1 | 49.2 | 65.1 | 64.3
  Week 1: >=50% reduction | 25.0 | 40.5 | 33.3 | 45.3 | 51.2
  Week 1: >=70% reduction | 13.9 | 23.0 | 23.8 | 27.9 | 33.3
  Week 1: >=90% reduction | 8.3 | 9.5 | 11.1 | 5.8 | 14.3
  Week 2: >=30% reduction | 48.6 | 63.5 | 57.1 | 61.6 | 54.8
  Week 2: >=50% reduction | 30.6 | 52.7 | 44.4 | 38.4 | 39.3
  Week 2: >=70% reduction | 18.1 | 36.5 | 30.2 | 27.9 | 20.2
  Week 2: >=90% reduction | 8.3 | 17.6 | 15.9 | 14.0 | 6.0
  Week 4: >=30% reduction | 56.9 | 66.2 | 65.1 | 66.3 | 66.7
  Week 4: >=50% reduction | 31.9 | 55.4 | 54.0 | 53.5 | 53.6
  Week 4: >=70% reduction | 19.4 | 44.6 | 34.9 | 43.0 | 32.1
  Week 4: >=90% reduction | 5.6 | 27.0 | 19.0 | 16.3 | 13.1
  Week 8: >=30% reduction | 59.7 | 62.2 | 68.3 | 69.8 | 71.4
  Week 8: >=50% reduction | 33.3 | 47.3 | 57.1 | 53.5 | 51.2
  Week 8: >=70% reduction | 16.7 | 40.5 | 42.9 | 38.4 | 29.8
  Week 8: >=90% reduction | 4.2 | 24.3 | 19.0 | 15.1 | 16.7
  Week 12: >=30% reduction | 61.1 | 62.2 | 68.3 | 69.8 | 70.2
  Week 12: >=50% reduction | 34.7 | 45.9 | 57.1 | 53.5 | 51.2
  Week 12: >=70% reduction | 18.1 | 40.5 | 42.9 | 38.4 | 31.0
  Week 12: >=90% reduction | 4.2 | 24.3 | 19.0 | 14.0 | 17.9
  Week 16: >=30% reduction | 61.1 | 60.8 | 68.3 | 69.8 | 70.2
  Week 16: >=50% reduction | 33.3 | 45.9 | 57.1 | 53.5 | 52.4
  Week 16: >=70% reduction | 18.1 | 40.5 | 41.3 | 38.4 | 31.0
  Week 16: >=90% reduction | 4.2 | 24.3 | 17.5 | 14.0 | 17.9

9. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Pain Subscale Score at Weeks 1, 2, 4, 8, 12, and 16
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index knee in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a NRS of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain. Participants with specified reduction (as percent) from baseline at Week 16 are reported.
Time Frame: Weeks 1, 2, 4, 8, 12, 16
Population: ITT population. LOCF method was used to impute missing values. Results for Week 1, 2, 4, 8 and 12 were not reported because analysis was not performed as per change in planned analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
Participants
  Week 16: Greater than 0% reduction | 63 | 69 | 57 | 77 | 78
  Week 16: >=10% reduction | 57 | 64 | 53 | 72 | 73
  Week 16: >=20% reduction | 50 | 56 | 47 | 65 | 65
  Week 16: >=30% reduction | 44 | 45 | 43 | 60 | 59
  Week 16: >=40% reduction | 32 | 40 | 39 | 54 | 52
  Week 16: >=50% reduction | 24 | 34 | 36 | 46 | 44
  Week 16: >=60% reduction | 21 | 30 | 29 | 42 | 34
  Week 16: >=70% reduction | 13 | 30 | 26 | 33 | 26
  Week 16: >=80% reduction | 11 | 24 | 17 | 22 | 21
  Week 16: >=90% reduction | 3 | 18 | 11 | 12 | 15
  Week 16: 100% reduction | 1 | 8 | 3 | 5 | 8

10. Secondary Outcome: Number of Participants With Improvement of at Least 2 Points in Patient's Global Assessment (PGA) of Osteoarthritis
Description: Participants answered the question: "Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?" Participants responded by using a 5-point scale where 1 = very good (asymptomatic and no limitation of normal activities), 2 = good (mild symptoms and no limitation of normal activities), 3 = fair (moderate symptoms and limitation of some normal activities), 4 = poor (severe symptoms and inability to carry out most normal activities) and 5 = very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher score indicated severe condition. Improvement signifies a decrease of at least 2 points on the 5-point scale relative to baseline value.
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
Participants
  Week 1 | 11 | 17 | 12 | 21 | 24
  Week 2 | 10 | 23 | 15 | 23 | 10
  Week 4 | 9 | 24 | 20 | 25 | 18
  Week 8 | 13 | 22 | 16 | 27 | 23
  Week 12 | 14 | 21 | 16 | 27 | 24
  Week 16 | 14 | 21 | 15 | 27 | 24

11. Secondary Outcome: Change From Baseline in Average Pain Score in the Index Knee at Weeks 1, 2, 4, 8, 12 and 16
Description: Participants assessed average osteoarthritis pain in their knee in the past 24 hours on an 11-point NRS ranging from 0 (no pain) to 10 (worst pain). Higher score indicated greater pain. Baseline score was calculated as the mean of the scores over the 3 days in the initial pain assessment period and a weekly mean was calculated using the daily pain scores within each study week.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, and 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). LOCF method was used to impute missing values. Here 'overall number of participants analyzed' included those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 70 | 74 | 62 | 85 | 84
units on a scale
  Baseline | 7.12 (1.75) | 6.96 (1.97) | 6.72 (2.10) | 6.93 (1.76) | 6.44 (1.88)
  Change at Week 1 | -1.17 (1.93) | -1.36 (1.69) | -1.27 (1.73) | -1.93 (1.99) | -1.82 (1.96)
  Change at Week 2 | -1.74 (2.27) | -2.54 (2.25) | -2.23 (2.33) | -2.47 (2.62) | -1.78 (2.17)
  Change at Week 4 | -2.10 (2.30) | -2.85 (2.35) | -2.95 (2.41) | -3.12 (2.73) | -2.37 (2.25)
  Change at Week 8 | -2.27 (2.60) | -2.55 (2.47) | -2.85 (2.26) | -3.01 (2.63) | -2.34 (2.34)
  Change at Week 12 | -2.32 (2.59) | -2.48 (2.44) | -3.00 (2.43) | -3.00 (2.68) | -2.34 (2.29)
  Change at Week 16 | -2.33 (2.59) | -2.49 (2.45) | -2.93 (2.39) | -2.97 (2.65) | -2.33 (2.29)

12. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 1, 2, 4, 8, 12, and 16
Description: The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced in the index joint in the past 48 hours. It is calculated as the mean of the scores from the 2 individual questions scored on NRS of 0 to 10, with higher scores indicating more stiffness. Total score range for WOMAC stiffness subscale score is 0 to 10, where higher scores indicate more stiffness. Stiffness is defined as a sensation of decreased ease in movement of the knee.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Baseline | 7.19 (1.78) | 7.33 (2.20) | 7.26 (1.73) | 7.41 (1.59) | 6.99 (1.85)
  Change at Week 1 | -1.75 (1.92) | -2.78 (2.65) | -2.40 (2.44) | -3.18 (2.65) | -3.24 (2.70)
  Change at Week 2 | -2.05 (2.11) | -3.38 (2.81) | -3.10 (2.71) | -3.38 (2.74) | -2.64 (2.61)
  Change at Week 4 | -2.17 (2.19) | -3.61 (3.05) | -3.52 (2.70) | -3.85 (2.82) | -3.38 (2.72)
  Change at Week 8 | -2.15 (2.04) | -3.32 (3.18) | -3.52 (2.68) | -3.87 (2.89) | -3.32 (2.66)
  Change at Week 12 | -2.19 (2.03) | -3.30 (3.19) | -3.52 (2.69) | -3.86 (2.87) | -3.36 (2.71)
  Change at Week 16 | -2.17 (2.03) | -3.30 (3.20) | -3.47 (2.64) | -3.87 (2.87) | -3.37 (2.69)

13. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 1, 2, 4, 8, 12, and 16
Description: WOMAC: self-administered, disease-specific 24-item questionnaire, which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores. WOMAC pain, physical function and stiffness subscale and average score ranges from 0 to 10, where higher score indicates worse response.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Baseline | 7.17 (1.44) | 7.43 (1.58) | 7.26 (1.44) | 7.35 (1.27) | 6.99 (1.30)
  Change at Week 1 | -1.88 (2.04) | -2.89 (2.36) | -2.43 (2.25) | -3.15 (2.37) | -3.21 (2.48)
  Change at Week 2 | -2.18 (2.01) | -3.48 (2.59) | -3.07 (2.55) | -3.19 (2.50) | -2.56 (2.37)
  Change at Week 4 | -2.39 (2.00) | -3.78 (2.72) | -3.46 (2.49) | -3.77 (2.60) | -3.37 (2.36)
  Change at Week 8 | -2.40 (1.88) | -3.52 (2.79) | -3.54 (2.50) | -3.76 (2.59) | -3.34 (2.27)
  Change at Week 12 | -2.45 (1.90) | -3.50 (2.79) | -3.54 (2.53) | -3.75 (2.58) | -3.38 (2.31)
  Change at Week 16 | -2.44 (1.90) | -3.49 (2.81) | -3.49 (2.47) | -3.75 (2.58) | -3.39 (2.30)

14. Secondary Outcome: Change From Baseline For Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 1, 2, 4, 8, 12, and 16
Description: Participants answered: "How much pain have you had when walking on a flat surface?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Baseline | 7.28 (1.69) | 7.73 (1.74) | 7.43 (1.71) | 7.41 (1.58) | 7.24 (1.68)
  Change at Week 1 | -2.01 (2.76) | -3.14 (2.54) | -2.67 (2.74) | -3.30 (2.67) | -3.40 (2.83)
  Change at Week 2 | -2.40 (2.75) | -3.82 (2.82) | -3.29 (2.77) | -3.26 (2.81) | -2.75 (2.82)
  Change at Week 4 | -2.68 (2.63) | -4.20 (2.94) | -3.60 (2.67) | -3.91 (2.89) | -3.64 (2.56)
  Change at Week 8 | -2.51 (2.49) | -4.01 (2.94) | -3.84 (2.71) | -3.85 (2.85) | -3.62 (2.50)
  Change at Week 12 | -2.57 (2.53) | -3.99 (2.94) | -3.84 (2.74) | -3.84 (2.84) | -3.64 (2.54)
  Change at Week 16 | -2.56 (2.53) | -3.99 (2.96) | -3.83 (2.72) | -3.85 (2.83) | -3.65 (2.54)

15. Secondary Outcome: Change From Baseline For Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Down Stairs at Weeks 1, 2, 4, 8, 12, and 16
Description: Participants answered: "How much pain have you had when going up or down stairs?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain. Higher score indicated greater pain.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
units on a scale
  Baseline | 8.50 (1.39) | 8.65 (1.34) | 8.44 (1.17) | 8.40 (1.33) | 8.25 (1.26)
  Change at Week 1 | -2.21 (2.75) | -3.14 (2.56) | -2.71 (2.69) | -3.30 (2.59) | -3.45 (2.95)
  Change at Week 2 | -2.74 (2.72) | -3.93 (2.93) | -3.54 (2.82) | -3.50 (2.99) | -2.95 (2.83)
  Change at Week 4 | -2.92 (2.69) | -4.36 (3.00) | -3.76 (2.84) | -4.08 (3.02) | -3.89 (2.58)
  Change at Week 8 | -2.85 (2.57) | -4.03 (3.06) | -3.98 (2.76) | -3.98 (2.93) | -3.86 (2.60)
  Change at Week 12 | -2.93 (2.61) | -4.00 (3.04) | -3.98 (2.78) | -3.98 (2.94) | -3.89 (2.64)
  Change at Week 16 | -2.92 (2.60) | -3.96 (3.08) | -3.94 (2.73) | -3.99 (2.94) | -3.92 (2.62)

16. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 16
Description: SF-36v2 is a standardized self-administered survey evaluating 8 aspects/domains of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The total score for each domain is scaled 0-100 (100 = highest level of functioning).
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 71 | 73 | 62 | 86 | 84
units on a scale
  Baseline: General Health Score | 66.01 (18.38) | 66.81 (20.54) | 68.73 (17.95) | 65.72 (19.98) | 65.02 (19.42)
  Baseline: Physical Function Score | 34.30 (23.80) | 32.05 (20.80) | 30.63 (18.07) | 38.55 (23.58) | 37.35 (21.80)
  Baseline: Role Physical Score | 40.85 (27.57) | 42.64 (27.68) | 39.42 (23.07) | 47.31 (27.70) | 49.03 (27.03)
  Baseline: Bodily Pain Score | 34.18 (19.25) | 32.85 (16.97) | 34.10 (17.02) | 33.70 (19.80) | 36.31 (18.06)
  Baseline: Vitality Score | 50.62 (20.97) | 52.91 (21.98) | 55.04 (18.35) | 51.74 (20.49) | 50.45 (19.97)
  Baseline: Social Function Score | 64.96 (30.95) | 69.69 (26.59) | 72.18 (24.94) | 65.41 (28.42) | 69.79 (25.61)
  Baseline: Role Emotional Score | 67.72 (31.81) | 73.63 (32.36) | 73.25 (29.99) | 73.45 (30.85) | 73.31 (28.22)
  Baseline: Mental Health Score | 72.89 (20.03) | 73.90 (19.10) | 77.82 (16.59) | 75.41 (17.41) | 75.77 (16.84)
  Change at Week 16: General Health Score | 0.07 (0.59) | -0.48 (2.91) | -0.08 (0.64) | 0.00 (0.00) | 0.44 (4.04)
  Change at Week 16: Physical Function Score | 0.35 (2.97) | -0.21 (4.75) | 0.48 (3.81) | 0.35 (3.23) | 0.06 (0.55)
  Change at Week 16: Role Physical Score | 0.26 (2.23) | -0.77 (9.99) | 0.20 (1.59) | 0.00 (0.00) | 0.22 (2.05)
  Change at Week 16: Bodily Pain Score | 0.30 (2.49) | -0.29 (2.34) | 0.31 (2.41) | 0.00 (0.00) | 0.36 (3.27)
  Change at Week 16: Vitality Score | 0.18 (1.48) | -0.43 (3.66) | -0.40 (3.18) | 0.07 (0.67) | 0.22 (2.05)
  Change at Week 16: Social Function Score | 0.18 (1.48) | -0.34 (2.93) | 0.60 (4.76) | 0.29 (2.70) | 0.30 (2.73)
  Change at Week 16: Role Emotional Score | 0.00 (0.00) | 0.68 (5.85) | 0.13 (1.06) | 0.29 (2.70) | 0.10 (0.91)
  Change at Week 16: Mental Health Score | 0.00 (0.00) | 0.14 (1.17) | -0.56 (4.45) | 0.23 (2.16) | -0.18 (1.64)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 16
Description: SF-36v2: standardized self-administered survey evaluating 8 aspects of functional health and wellbeing (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health). Total score for each aspect were scaled 0-100 (100=highest level of functioning). For obtaining physical and mental component scores, z-score for each scale=(observed score - mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 71 | 73 | 62 | 86 | 84
z-score
  Baseline: Physical Component Score | -1.78 (0.81) | -1.86 (0.79) | -1.93 (0.70) | -1.71 (0.88) | -1.68 (0.82)
  Baseline: Mental Component Score | 0.03 (1.25) | 0.27 (1.23) | 0.44 (1.11) | 0.16 (1.17) | 0.19 (1.08)
  Change at Week 16: Physical Component Score | 0.01 (0.12) | -0.03 (0.26) | 0.02 (0.15) | 0.00 (0.01) | 0.02 (0.14)
  Change at Week 16: Mental Component Score | -0.00 (0.02) | 0.02 (0.09) | -0.02 (0.13) | 0.01 (0.12) | -0.00 (0.00)

18. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy for participants who discontinued due to lack of efficacy was reported.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of intravenous or subcutaneous study medication (either tanezumab or matching placebo). Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 4 | 3 | 1 | 0 | 4
days | 14.0 [8 to 25] | 29.0 [8 to 57] | 8.0 [8 to 8] |  | 16.5 [8 to 21]

19. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication. Incidence of rescue medication use is calculated as any use of rescue medication during the study week in question.
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: ITT population. LOCF method was used to impute missing values. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 71 | 73 | 59 | 82 | 81
percentage of participants
  Week 1: number analyzed (Participants) | 70 | 73 | 57 | 81 | 80
  Week 1 | 70.0 | 54.8 | 57.9 | 53.1 | 50.0
  Week 2: number analyzed (Participants) | 71 | 73 | 59 | 82 | 80
  Week 2 | 56.3 | 47.9 | 52.5 | 57.3 | 55.0
  Week 4 | 43.7 | 38.4 | 39.0 | 40.2 | 37.0
  Week 8 | 45.1 | 30.1 | 40.7 | 35.4 | 42.0
  Week 12 | 43.7 | 28.8 | 39.0 | 35.4 | 39.5
  Week 16 | 43.7 | 28.8 | 39.0 | 35.4 | 39.5

20. Secondary Outcome: Duration of Rescue Medication Use
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication. Duration of rescue medication use is calculated as the number of study days per week when any rescue medication was taken.
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 71 | 73 | 59 | 82 | 81
days/week
  Week 1: number analyzed (Participants) | 70 | 73 | 57 | 81 | 80
  Week 1 | 2.2 (2.25) | 1.8 (2.14) | 1.7 (2.01) | 1.6 (2.07) | 1.5 (2.13)
  Week 2: number analyzed (Participants) | 71 | 73 | 59 | 82 | 80
  Week 2 | 2.0 (2.27) | 1.3 (1.88) | 1.7 (2.06) | 1.5 (1.72) | 1.7 (2.15)
  Week 4 | 1.6 (2.41) | 1.0 (1.63) | 1.2 (2.01) | 1.0 (1.82) | 1.4 (2.33)
  Week 8 | 1.6 (2.41) | 0.8 (1.48) | 1.5 (2.32) | 0.8 (1.61) | 1.5 (2.33)
  Week 12 | 1.5 (2.32) | 0.8 (1.53) | 1.4 (2.29) | 0.8 (1.69) | 1.4 (2.33)
  Week 16 | 1.5 (2.32) | 0.8 (1.53) | 1.4 (2.29) | 0.8 (1.69) | 1.4 (2.33)

21. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 3000 mg per day up to 3 days per week could be taken as rescue medication. The amount of rescue medication taken is the total dose (in mg) of acetaminophen rescue medication over the study week in question.
Time Frame: Weeks 1, 2, 4, 8, 12, and 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 71 | 73 | 59 | 82 | 81
mg/week
  Week 1: number analyzed (Participants) | 70 | 73 | 57 | 81 | 80
  Week 1 | 3128.57 (3529.06) | 2609.59 (3737.24) | 2324.56 (3291.62) | 2425.93 (3976.58) | 1631.25 (2616.58)
  Week 2: number analyzed (Participants) | 71 | 73 | 59 | 82 | 80
  Week 2 | 3077.46 (4623.42) | 1753.42 (3210.36) | 2440.68 (3312.83) | 2189.02 (3864.72) | 2425.00 (3693.22)
  Week 4 | 2556.34 (4842.93) | 1239.73 (2691.43) | 1889.83 (4100.11) | 1445.12 (2946.02) | 1716.05 (3534.60)
  Week 8 | 2464.79 (4729.33) | 1047.95 (2636.77) | 2042.37 (4175.35) | 981.71 (2028.26) | 1777.78 (3280.62)
  Week 12 | 2140.85 (4297.16) | 1061.64 (2658.77) | 1940.68 (4132.59) | 951.22 (1888.25) | 1654.32 (3242.92)
  Week 16 | 2140.85 (4297.16) | 1061.64 (2658.77) | 1940.68 (4132.59) | 951.22 (1888.25) | 1654.32 (3242.92)

22. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 112 days after last dose of study treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
Participants
  AEs | 37 | 35 | 31 | 36 | 44
  SAEs | 2 | 2 | 0 | 0 | 1

23. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Findings
Description: Laboratory examination included blood chemistry, hematology and urinalysis. Reported results include abnormal laboratory findings without regard to baseline abnormality.
Time Frame: Day 1 up to Week 24
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 68 | 71 | 61 | 82 | 83
Participants | 56 | 48 | 44 | 61 | 60

24. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Following parameters were analyzed for ECG abnormality: PR interval, QRS interval, QT interval, QT interval corrected using the Fridericia's formula (QTcF), QT interval corrected using the Bazett's formula (QTcB), RR interval and heart rate (HR). Number of participants with clinically significant abnormal ECG findings reported as adverse events were presented.
Time Frame: Baseline up to Week 24
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 70 | 73 | 62 | 84 | 84
Participants | 0 | 1 | 1 | 0 | 1

25. Other Pre Specified Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16, and 24
Description: The NIS constitutes the sum of 37 standard items of neuromuscular examination used to assess the muscle strength, reflexes and sensation. Each item is scored separately for left and right sides. Components of muscle weakness (24 items) are scored on a scale from 0 (normal) to 4 (paralysis), with higher score = more weakness; components of reflexes and sensation (13 items) scored on a scale with 0 = normal, 1 = decreased or 2 = absent. Total NIS score range 0-244 with higher score = more impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 72 | 63 | 85 | 84
units on a scale
  Baseline | 1.06 (3.13) | 1.53 (5.09) | 0.86 (2.40) | 0.75 (2.69) | 1.71 (3.85)
  Change at Week 2: number analyzed (Participants) | 66 | 68 | 61 | 80 | 73
  Change at Week 2 | -0.09 (2.20) | -0.26 (1.79) | -0.13 (0.72) | -0.08 (1.97) | -0.36 (2.17)
  Change at Week 4: number analyzed (Participants) | 70 | 70 | 62 | 82 | 83
  Change at Week 4 | 0.11 (1.31) | -0.14 (2.22) | -0.19 (0.87) | -0.22 (1.51) | 0.14 (3.14)
  Change at Week 8: number analyzed (Participants) | 70 | 70 | 62 | 82 | 83
  Change at Week 8 | -0.07 (1.60) | -0.14 (2.34) | -0.26 (0.99) | -0.20 (1.59) | -0.39 (2.45)
  Change at Week 12: number analyzed (Participants) | 70 | 71 | 62 | 82 | 83
  Change at Week 12 | -0.10 (1.47) | -0.27 (2.07) | -0.32 (1.32) | -0.40 (2.34) | -0.81 (2.80)
  Change at Week 16: number analyzed (Participants) | 70 | 71 | 62 | 82 | 84
  Change at Week 16 | -0.16 (1.15) | -0.63 (2.60) | -0.23 (1.26) | -0.33 (1.65) | -0.62 (2.18)
  Change at Week 24: number analyzed (Participants) | 70 | 71 | 62 | 82 | 84
  Change at Week 24 | -0.19 (2.02) | -0.86 (3.05) | -0.55 (1.53) | -0.52 (2.01) | -0.90 (2.34)

26. Other Pre Specified Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA). Same participant may have positive ADA result at more than 1 time point.
Time Frame: Baseline, Weeks 8, 16, 24 or Early Termination
Population: ITT population. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure at any time point and 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 75 | 66 | 87 | 85
Participants
  Baseline: number analyzed (Participants) | 68 | 57 | 79 | 76
  Baseline | 0 | 0 | 1 | 0
  Week 8: number analyzed (Participants) | 59 | 52 | 75 | 68
  Week 8 | 1 | 0 | 1 | 0
  Week 16: number analyzed (Participants) | 7 | 5 | 8 | 6
  Week 16 | 0 | 0 | 0 | 0
  Week 24 (End of treatment): number analyzed (Participants) | 62 | 59 | 71 | 73
  Week 24 (End of treatment) | 1 | 3 | 1 | 1

27. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included examination of following sites in addition to general examination: abdomen, ears, extremities, eyes, head, heart, musculoskeletal, neck, nose, skin, throat, lungs and thyroid.
Time Frame: Baseline up to Week 24
Population: Data was not summarized separately and any clinically significant abnormality in physical finding was reported as an adverse event in this study.
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Other Pre Specified Outcome: Number of Participants With Clinically Significant Abnormality in Vital Signs
Description: Following parameters were analyzed for examination of vital signs: body temperature, blood pressure, pulse rate and respiratory rate. Number of participants with clinically significant abnormality in vital signs reported as adverse events were presented.
Time Frame: Baseline to Week 24
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 73 | 63 | 86 | 84
Participants | 1 | 0 | 1 | 1 | 0

29. Other Pre Specified Outcome: Number of Participants With Injection and Infusion Site Reactions
Description: The injection and infusion site reactions were assessed based on presence of erythema (redness), induration (swelling), ecchymosis (bruising), pruritus (itching) and pain that occurred after administration of subcutaneous injection or intravenous infusion.
Time Frame: Baseline, Weeks 1, 2, 4, 8, 12, 16, and 24
Population: ITT population. Here 'overall number of participants analyzed' signifies those participants who were evaluable for this measure and 'number analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 72 | 63 | 85 | 84
Participants
  Baseline: Injection site: number analyzed (Participants) | 71 | 72 | 63 | 85 | 84
  Baseline: Injection site | 1 | 2 | 0 | 1 | 1
  Baseline: Infusion site | 1 | 2 | 1 | 1 | 0
  Week 1: Injection site: number analyzed (Participants) | 66 | 72 | 60 | 81 | 81
  Week 1: Injection site | 1 | 0 | 0 | 2 | 1
  Week 1: Infusion site: number analyzed (Participants) | 67 | 72 | 60 | 81 | 81
  Week 1: Infusion site | 1 | 0 | 0 | 0 | 2
  Week 2: Injection site: number analyzed (Participants) | 64 | 69 | 59 | 81 | 76
  Week 2: Injection site | 0 | 0 | 0 | 0 | 1
  Week 2: Infusion site: number analyzed (Participants) | 65 | 69 | 59 | 81 | 76
  Week 2: Infusion site | 0 | 0 | 0 | 0 | 0
  Week 4: Injection site: number analyzed (Participants) | 60 | 68 | 58 | 81 | 77
  Week 4: Injection site | 0 | 0 | 0 | 0 | 0
  Week 4: Infusion site: number analyzed (Participants) | 61 | 68 | 58 | 81 | 77
  Week 4: Infusion site | 0 | 0 | 0 | 0 | 0
  Week 8: Injection site: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7
  Week 8: Injection site | 0 | 0 | 0 | 0 | 0
  Week 8: Infusion site: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7
  Week 8: Infusion site | 0 | 0 | 0 | 0 | 0
  Week 12: Injection site: number analyzed (Participants) | 8 | 8 | 7 | 9 | 7
  Week 12: Injection site | 0 | 0 | 0 | 0 | 0
  Week 12: Infusion site: number analyzed (Participants) | 8 | 8 | 7 | 9 | 7
  Week 12: Infusion site | 0 | 0 | 0 | 0 | 0
  Week 16: Injection site: number analyzed (Participants) | 4 | 8 | 5 | 8 | 8
  Week 16: Injection site | 0 | 0 | 0 | 0 | 0
  Week 16: Infusion site: number analyzed (Participants) | 4 | 8 | 5 | 8 | 8
  Week 16: Infusion site | 0 | 0 | 0 | 0 | 0
  Week 24: Injection site: number analyzed (Participants) | 5 | 7 | 5 | 8 | 7
  Week 24: Injection site | 0 | 0 | 0 | 0 | 0
  Week 24: Infusion site: number analyzed (Participants) | 5 | 7 | 5 | 8 | 7
  Week 24: Infusion site | 0 | 0 | 0 | 0 | 0

30. Other Pre Specified Outcome: Plasma Tanezumab Concentration
Time Frame: Baseline (pre-dose), Weeks 1, 2, 4, 8 (pre-dose), 12, 16, 24 or End of treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 69 | 60 | 82 | 80
nanogram per milliliter (ng/mL)
  Baseline: pre-dose: number analyzed (Participants) | 68 | 58 | 78 | 80
  Baseline: pre-dose | 12.65 (36.610) | 14.43 (45.560) | 30.90 (81.647) | 138.5 (820.35)
  Week 1: number analyzed (Participants) | 69 | 60 | 81 | 79
  Week 1 | 265.7 (132.17) | 480.7 (249.53) | 1015 (429.96) | 1700 (874.30)
  Week 2: number analyzed (Participants) | 67 | 56 | 82 | 76
  Week 2 | 270.2 (110.93) | 486.3 (160.85) | 1012 (350.47) | 1378 (772.25)
  Week 4: number analyzed (Participants) | 64 | 56 | 77 | 71
  Week 4 | 207.4 (95.228) | 371.8 (185.63) | 791.1 (228.97) | 887.5 (280.47)
  Week 8: pre-dose: number analyzed (Participants) | 59 | 53 | 74 | 70
  Week 8: pre-dose | 81.51 (59.632) | 158.1 (89.087) | 370.2 (176.99) | 428.1 (213.49)
  Week 12: number analyzed (Participants) | 53 | 53 | 67 | 64
  Week 12 | 52.55 (92.620) | 88.13 (150.90) | 323.8 (349.02) | 304.8 (286.23)
  Week 16: number analyzed (Participants) | 7 | 5 | 8 | 6
  Week 16 | 99.73 (70.613) | 257.0 (298.20) | 628.6 (244.38) | 501.7 (218.74)
  Week 24 (End of treatment): number analyzed (Participants) | 62 | 59 | 62 | 73
  Week 24 (End of treatment) | 17.58 (38.959) | 58.57 (142.04) | 113.2 (139.49) | 264.2 (960.42)

31. Other Pre Specified Outcome: Total and Free Nerve Growth Factor (NGF) Concentration
Description: Serum samples were analyzed for determining total and free (unbound) NGF concentration. Total NGF was analyzed using a validated, sensitive and specific immunoaffinity enrichment liquid chromatography tandem mass spectrometric (IA/LC/MS/MS) method and free (unbound) NGF was analyzed using a validated, sensitive, and specific electrochemiluminescence (ECL) ligand binding assay.
Time Frame: Baseline (pre-dose), Weeks 1, 2, 4, 8 (pre-dose), 12, 16, and 24 or End of treatment
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 66 | 69 | 60 | 82 | 80
picogram per milliliter (pg/mL)
  Baseline (pre-dose): Total NGF: number analyzed (Participants) | 43 | 35 | 41 | 54 | 55
  Baseline (pre-dose): Total NGF | 34.9 (10.1) | 44.6 (41.8) | 79.2 (276) | 35.1 (8.7) | 32.7 (9.2)
  Baseline (pre-dose): Free NGF: number analyzed (Participants) | 66 | 69 | 58 | 79 | 80
  Baseline (pre-dose): Free NGF | 1.7 (0.9) | 1.8 (1.0) | 1.6 (0.8) | 1.5 (0.7) | 1.5 (0.8)
  Week 1: Total NGF: number analyzed (Participants) | 43 | 35 | 41 | 54 | 55
  Week 1: Total NGF | 71.3 (232) | 742 (302) | 941 (419) | 1196 (452) | 1432 (477)
  Week 1: Free NGF: number analyzed (Participants) | 63 | 68 | 60 | 78 | 77
  Week 1: Free NGF | 1.6 (1.2) | 1.1 (1.1) | 0.9 (2.1) | 0.2 (0.6) | 0.1 (0.4)
  Week 2: Total NGF: number analyzed (Participants) | 43 | 66 | 56 | 82 | 74
  Week 2: Total NGF | 35.0 (13.8) | 1202 (400) | 1497 (532) | 1867 (588) | 2149 (601)
  Week 2: Free NGF: number analyzed (Participants) | 64 | 67 | 56 | 82 | 74
  Week 2: Free NGF | 1.7 (0.7) | 2.5 (1.4) | 2.1 (1.4) | 0.8 (1.0) | 0.8 (1.2)
  Week 4: Total NGF: number analyzed (Participants) | 42 | 64 | 55 | 76 | 71
  Week 4: Total NGF | 35.5 (13.4) | 1596 (542) | 2108 (1129) | 2554 (828) | 2629 (750)
  Week 4: Free NGF: number analyzed (Participants) | 62 | 64 | 55 | 77 | 71
  Week 4: Free NGF | 1.7 (1.0) | 3.3 (1.5) | 3.4 (1.4) | 2.5 (1.3) | 2.7 (1.4)
  Week 8 (pre-dose): Total NGF: number analyzed (Participants) | 40 | 57 | 53 | 75 | 70
  Week 8 (pre-dose): Total NGF | 35.7 (12.8) | 1388 (606) | 1867 (890) | 2544 (869) | 2724 (931)
  Week 8 (pre-dose): Free NGF: number analyzed (Participants) | 55 | 58 | 53 | 74 | 70
  Week 8 (pre-dose): Free NGF | 1.6 (0.8) | 2.3 (1.3) | 3.1 (1.4) | 4.5 (2.5) | 4.7 (1.9)
  Week 12: Total NGF: number analyzed (Participants) | 32 | 52 | 52 | 66 | 64
  Week 12: Total NGF | 33.7 (13.1) | 798 (768) | 1216 (751) | 2253 (1024) | 2521 (1166)
  Week 12: Free NGF: number analyzed (Participants) | 50 | 54 | 53 | 67 | 64
  Week 12: Free NGF | 1.7 (0.9) | 1.4 (1.3) | 1.9 (1.6) | 3.1 (1.8) | 3.5 (1.8)
  Week 16: Total NGF: number analyzed (Participants) | 4 | 7 | 5 | 8 | 6
  Week 16: Total NGF | 35.2 (10.1) | 1900 (1428) | 1206 (830) | 3320 (502) | 4082 (1940)
  Week 16: Free NGF: number analyzed (Participants) | 6 | 7 | 5 | 8 | 6
  Week 16: Free NGF | 2.0 (0.7) | 1.9 (1.2) | 3.7 (4.1) | 5.9 (4.3) | 5.3 (1.5)
  Week 24 (End of treatment): Total NGF: number analyzed (Participants) | 38 | 54 | 51 | 71 | 71
  Week 24 (End of treatment): Total NGF | 31.7 (10.9) | 251 (323) | 489 (634) | 1114 (737) | 1445 (997)
  Week 24 (End of treatment): Free NGF: number analyzed (Participants) | 57 | 62 | 59 | 71 | 72
  Week 24 (End of treatment): Free NGF | 1.6 (1.0) | 1.5 (0.9) | 1.5 (1.0) | 2.1 (2.0) | 2.0 (1.5)

32. Other Pre Specified Outcome: Number of Participants With Intravenous or Subcutaneous Doses of Study Medication
Description: Number of participants were reported based on the maximum number of intravenous or subcutaneous doses of either tanezumab or placebo received.
Time Frame: Baseline up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Number analyzed (Participants) | 72 | 74 | 63 | 86 | 84
Participants
  1 dose | 65 | 67 | 56 | 78 | 77
  2 doses | 7 | 7 | 7 | 8 | 7

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Tanezumab 2.5 mg Subcutaneous Injection | Tanezumab 5 mg Subcutaneous Injection | Tanezumab 10 mg Subcutaneous Injection | Tanezumab 10 mg Intravenous Infusion
Serious Adverse Events (participants affected / at risk) | 2/72 | 2/74 | 0/63 | 0/86 | 1/84
Other Adverse Events (participants affected / at risk) | 26/72 | 24/74 | 22/63 | 29/86 | 31/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Tanezumab 2.5 mg Subcutaneous Injection (N=74) | Tanezumab 5 mg Subcutaneous Injection (N=63) | Tanezumab 10 mg Subcutaneous Injection (N=86) | Tanezumab 10 mg Intravenous Infusion (N=84)
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Tanezumab 2.5 mg Subcutaneous Injection (N=74) | Tanezumab 5 mg Subcutaneous Injection (N=63) | Tanezumab 10 mg Subcutaneous Injection (N=86) | Tanezumab 10 mg Intravenous Infusion (N=84)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 2
Infusion site reaction (General disorders) | 1 | 2 | 1 | 1 | 2
Injection site reaction (General disorders) | 2 | 2 | 0 | 4 | 3
Oedema peripheral (General disorders) | 0 | 1 | 3 | 4 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 7 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 4 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 5 | 0 | 5 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 6 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 6 | 6
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to United States Food and Drug Administration (FDA) imposed clinical hold, enrollment was stopped prematurely and, therefore, was insufficient to yield adequate power to fulfill the primary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.